CLINICAL TRIAL: NCT01399853
Title: A Phase II Clinical Trial for Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT005
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Immunogenicity; Safety
Keywords: immunogenicity; safety; inactivated EV71 vaccine
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 160U /0.5ml in children (from 12 to 36 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 160U /0.5ml in 120 children aged 12-36 months old on day0,28
  Interventions: Biological: 160U /0.5ml EV71 Vaccine
- 320U /0.5ml in children (from 12 to 36 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 120 children aged 12-36 months old on day0,28
  Interventions: Biological: 320U /0.5ml EV71 vaccine
- 640U /0.5ml in children (from 12 to 36 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 120 children aged 12-36 months old on day0,28
  Interventions: Biological: 640U /0.5ml EV71 vaccine
- (without adjuvant) 640U /0.5ml in children (12-36months) (Experimental): inactivated vaccine(vero cell) against EV71 of (without adjuvant) 640U /0.5ml in 120 children aged 12-36 months old on day0,28
  Interventions: Biological: (without adjuvant) 640U /0.5ml
- 160U /0.5ml in infants (from 6 to 11 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 160U /0.5ml in 120 infants aged 6-11 months old on day0,28
  Interventions: Biological: 160U /0.5ml EV71 Vaccine
- 320U /0.5ml in infants (from 6 to 11 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 120 infants aged 6-11 months old on day0,28
  Interventions: Biological: 320U /0.5ml EV71 vaccine
- 640U /0.5ml in infants (from 6 to 11 months old) (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 120 infants aged 6-11 months old on day0,28
  Interventions: Biological: 640U /0.5ml EV71 vaccine
- (without adjuvant) 640U /0.5ml in infants (from 6 to 11 months (Experimental): inactivated vaccine(vero cell) against EV71 of (without adjuvant) 640U /0.5ml in 120 infants aged 6-11 months old on day0,28
  Interventions: Biological: (without adjuvant) 640U /0.5ml
- 0/0.5ml placebo in children (from 12 to 36 months old) (Placebo Comparator): 0/0.5ml placebo in 120 children aged 12-36 months old on day0,28
  Interventions: Biological: 0/0.5ml placebo
- 0/0.5ml placebo in infants (from 6 to 11 months old) (Placebo Comparator): 0/0.5ml placebo in 120 infants aged 6-11 months old on day0,28
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: 160U /0.5ml EV71 Vaccine — inactivated vaccine (vero cell) against EV71 of 160U /0.5ml, two doses, 28 days interval
  Arms: 160U /0.5ml in children (from 12 to 36 months old); 160U /0.5ml in infants (from 6 to 11 months old)
Biological: 320U /0.5ml EV71 vaccine — inactivated vaccine(vero cell) against EV71 of 320U /0.5ml, two doses, 28 days interval
  Arms: 320U /0.5ml in children (from 12 to 36 months old); 320U /0.5ml in infants (from 6 to 11 months old)
Biological: 640U /0.5ml EV71 vaccine — inactivated vaccine (vero cell) against EV71 of 640U /0.5ml, two doses, 28 days interval
  Arms: 640U /0.5ml in children (from 12 to 36 months old); 640U /0.5ml in infants (from 6 to 11 months old)
Biological: (without adjuvant) 640U /0.5ml — inactivated vaccine (vero cell) against EV71 of (without adjuvant) 640U /0.5ml, two doses, 28 days interval
  Arms: (without adjuvant) 640U /0.5ml in children (12-36months); (without adjuvant) 640U /0.5ml in infants (from 6 to 11 months
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, 28 days interval
  Arms: 0/0.5ml placebo in children (from 12 to 36 months old); 0/0.5ml placebo in infants (from 6 to 11 months old)

SUMMARY:
Hand, foot, and mouth disease (HFMD) is a common viral illness in infants and children caused by viruses that belong to the enterovirus genus of the picornavirus family. Although most HFMD cases do not result in serious complications, outbreaks of HFMD caused by enterovirus 71 (EV71) can present with a high rate of neurological complications, including meningoencephalitis, pulmonary complications, and can even cause infant death. HFMD caused by EV71 has become a major emerging infectious disease in Asia and the highly pathogenic potential of EV71 clearly requires the attention of world medical community.

The phase I study of inactivated vaccine (vero cell) against EV71 has completed last month in Jiangsu Province in China. The data from the phase I study suggested that the inactivated EV71 vaccine had a clinically acceptable safety and good immunogenicity for healthy Chinese children and infants. In order to provide more evidence for the immunogenicity of the vaccine, to further explore the probable immunizing dose and the safety profile of this vaccine, a phase II clinical trial is planed to conduct.

ELIGIBILITY:
Inclusion Criteria:

For children group (aged from 12-36 months):

* Healthy children aged from 12 to 36 months old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

For infants group (aged from 6-11 months):

* Healthy infants aged from 6 to 11 months old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

For children group (aged from 12-36 months):

* Subject who has a medical history of HFMD
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Under the anti-TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

For infants group (aged from 6-11 months):

* Subject who has a medical history of HFMD
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Under the anti-TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second dose:

* Had any Grade 3 or Grade 4 adverse reaction within 7 days after first dose
* Any situation meet the exclusion criteria stated in the exclusion criteria for first dose
* Had any SAE related to first dose during the following-up of first dose
* Any condition that in the opinion of the investigator, or IRB

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The GMT of anti-EV71 antibodies in serum after first vaccination | 28 days after first vaccination
  to evaluate the GMT of anti-EV71 antibodies in serum 28 days after first vaccination
The GMT of anti-EV71 antibodies in serum after second vaccination | 28 days after second vaccination
  to evaluate the GMT of anti-EV71 antibodies in serum 28 days after second vaccination
Frequency of systemic and local adverse reactions after the first vaccination | 28 days after the first vaccination
  Frequency of systemic and local adverse reactions in healthy Children and infants following first doses of EV71 vaccine
Frequency of systemic and local adverse reactions after the second vaccination | 28 days after the second vaccination
  Frequency of systemic and local adverse reactions in healthy Children and infants following second doses of EV71 vaccine

SECONDARY OUTCOMES:
The seroconversion rate of anti-EV71 antibodies in serum after first vaccination | 28 days after first vaccination
  to evaluate the seroconversion rate of anti-EV71 antibodies in serum 28 days after first vaccination
The seroconversion rate of anti-EV71 antibodies in serum after second vaccination | 28 days after second vaccination
  to evaluate the seroconversion rate of anti-EV71 antibodies in serum 28 days after second vaccination
Frequency of adverse events and any SAE after the first vaccination | 28 days after the first vaccination
  Frequency of adverse events and any SAE in healthy Children and infants following first doses of EV71 vaccine
Frequency of adverse events and any SAE after the second vaccination | 28 days after the second vaccination
  Frequency of adverse events and any SAE in healthy Children and infants following second doses of EV71 vaccine
The clinical abnormality of hematological examination, blood biochemical test and urinalysis after first vaccination in children | 3 days after first vaccination
  to evaluate the clinical abnormality of hematological examination, blood biochemical test and urinalysis 3 days after first vaccination in children
The clinical abnormality of hematological examination, blood biochemical test and urinalysis after second vaccination in children | 3 days after second vaccination
  to evaluate the clinical abnormality of hematological examination, blood biochemical test and urinalysis 3 days after second vaccination in children
The persistence of immunogenicity of the EV71vaccine after two doses in children and infants | 6 months after blood collection at day 56
  to evaluate the persistence of immunogenicity of the EV71vaccine after two doses in children and infants 6 months after blood collection at day 56

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhu FC, Liang ZL, Li XL, Ge HM, Meng FY, Mao QY, Zhang YT, Hu YM, Zhang ZY, Li JX, Gao F, Chen QH, Zhu QY, Chu K, Wu X, Yao X, Guo HJ, Chen XQ, Liu P, Dong YY, Li FX, Shen XL, Wang JZ. Immunogenicity and safety of an enterovirus 71 vaccine in healthy Chinese children and infants: a randomised, double-blind, placebo-controlled phase 2 clinical trial. Lancet. 2013 Mar 23;381(9871):1037-45. doi: 10.1016/S0140-6736(12)61764-4. PMID 23352749